CLINICAL TRIAL: NCT07375992
Title: Music Therapy in Newly Diagnosed Glioblastoma After Chemoradiation Therapy (MELODY-GBM) J2556
Brief Title: Music Therapy in Newly Diagnosed Glioblastoma After Chemoradiation Therapy (MELODY-GBM)
Acronym: MELODY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Keep Punching Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J2556; IRB00493841 (Other: JHU IRB)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Feasibility Studies
Keywords: newly diagnosed; Glioblastoma; Music Therapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This study will assess the feasibility of Music Therapy in the high-risk, high-needs population of individuals newly diagnosed with GBM and undergoing standard of care adjuvant chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A- with Music Therapists (Experimental): Arm A of the study will involve individuals who are assigned to receive twice weekly music therapy sessions with a Music Therapist. These live sessions will be conducted virtually via a Johns Hopkins Compliance virtual platform (e.g., Zoom) each session will last 30 minutes. Participants will complete a total of 16 music therapy sessions, and the frequency is 2 sessions per week for 8 weeks. Participants will complete surveys measuring quality of life once each week.
  Interventions: Other: Music intervention
- Arm B- without Music Therapists (Experimental): Arm B of the study participants will meet with a music therapist to create a curated playlist. The participant will then listen independently to music therapy sessions twice a week for thirty minutes. Participants will complete a total of 16 music therapy sessions, and the frequency is 2 sessions per week for 8 weeks. Participants will complete surveys measuring quality of life once each week.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — Each GBM study participant in Arm A will receive two 30-minute live synchronous virtual music therapy sessions per week for a period of 8 weeks to be curated by a board-certified music therapist. Arm B participants will receive curated playlists of music created by a music therapist. Participants will then listen to the curated music playlists on the participant's own device twice per week.
  All participants will complete a total of 16 music therapy sessions, scheduled twice per week over 8 weeks. Each session will last approximately 30 minutes.

SUMMARY:
The Brain Cancer Program, in partnership with the Center for Music and Medicine at Johns Hopkins, will study whether music therapy is feasible in newly diagnosed GBM patients undergoing standard care.

DETAILED DESCRIPTION:
Virtually via Zoom, all participants will meet with Music Therapists to create playlists and learn how to complete surveys measuring quality of life.

Participants will be randomly assigned, half to each arm. Arm A will interact with Music Therapists and listen to music twice a week, then independently fill out quality of life questionnaires.

Arm B will listen to music independently twice a week, then independently fill out quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma
* Cognitive capacity to respond to surveys
* Access to computer and web access
* Ability to attend virtual music therapy sessions
* Audibly process music
* Proficient in English

Exclusion Criteria:

* Not planning to undergo standard of care radiation therapy and concurrent and adjuvant temozolomide.
* A life expectancy of less than 6 months.
* Concurrent use of any other standard or investigational agents (excepting tumor treating fields).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit adherence with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02-02 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of Music Therapy intervention for GBM patients | 6 months
  Determine success rate of the delivery of individualized virtual music therapy (MT) in participants undergoing standard of care treatment for newly diagnosed glioblastoma.

SECONDARY OUTCOMES:
Rate of survey completion | 2 years
  Rate of participants completing all surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Holdhoff, MD, Principal Investigator — Johns Hopkins -Sidney Kimmel Cancer Center; Grace Tobin, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- oncology- Broadway, Baltimore, Maryland, United States